CLINICAL TRIAL: NCT05305378
Title: Intraoperative Laser Speckle Contrast Imaging of Cerebral Blood Flow
Status: Completed | Type: Observational
Sponsor: Dynamic Light (Industry)
Collaborators: Barrow Neurological Institute (Other)
Responsible Party: Sponsor
Other Study IDs: LSCI-NSURG-03
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Aneurysm, AVM, Dural Arteriovenous Fistula, Glioma, Meningioma, Metastasis, Bypass
MeSH Terms: conditions — Aneurysm; Central Nervous System Vascular Malformations; Glioma; Meningioma; Neoplasm Metastasis | interventions — Laser Speckle Contrast Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Laser speckle contrast imaging (LSCI) — LSCI videos will be recorded intraoperatively in each patient before, during, and after ICGA in the same surgical field of view to guarantee comparability of the methods.

SUMMARY:
The purpose of the proposed study is to investigate the usefulness of laser speckle contrast imaging (LSCI) compared to indocyanine green angiography (ICGA). We will collect data from a wide variety of neurovascular surgical procedures to determine when the technology is the most clinically useful. The intraoperative LSCI system provides high resolution images of blood flow in real-time without tissue contact and without the need for an exogenous contrast agent. Further study is needed to gain a better understanding of the use of the technique during surgery, but initial results suggest that the ability to identify blood flow changes with immediate feedback to the surgeon could be a significant advantage during many procedures.

DETAILED DESCRIPTION:
Cerebral blood flow (CBF) is of paramount importance to human brain function, as the brain relies on a continuous blood supply to meet its energy needs. Blockage of a cerebral blood vessel during the course of surgery, even if transient and short-lived, may result in irreversible brain tissue damage (i.e. stroke) and loss of cortical function, if not identified quickly enough. During neurosurgery, vessel occlusion may occur either inadvertently or as a necessary part of the procedure, and yet current technologies do not adequately predict the consequences of such occlusion. Real-time CBF visualization during surgery could help neurosurgeons better understand the consequences of vascular occlusion events during surgery, recognize potential adverse complications, and thus prompt timely intervention to reduce the risk of stroke. The current standard for visualizing CBF during surgery is indocyanine green angiography (ICGA), which involves administering a bolus of fluorescent dye intravenously and imaging the wash-in of the dye to determine which vessels are perfused. Unfortunately, ICGA can only be used a few times during a surgery due to the need to inject a fluorescent dye, and provides only an instantaneous view of perfusion rather than a continuous view.

Patients will undergo standard craniotomy surgery. The surgical procedures will not be altered in any way by the proposed studies. As long as it is standard of care, neuromonitoring, intraoperative angiogram, and Indocyanine green angiography will be performed by the surgeon. LSCI imaging will be performed at the discretion of the surgeon following exposure of the cortex and will vary from patient to patient depending on the neurosurgical procedure. The LSCI measurements will not add any time to the surgery nor affect the normal operation of the neurosurgical microscope.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (18 years or older).
2. Size of craniotomy at least 2 cm.
3. Possibility of intraoperative ICGA.
4. Able to render written informed consent.
5. Women of child-bearing potential must have a negative pre-op pregnancy test.

Exclusion Criteria:

1. Patients unable to legally consent.
2. Patients with impaired cognitive function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seeking treatment at the Barrow Neurological Institute with pathologies that require a craniotomy of at least 2 cm in diameter.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Agreement of ICG and LSCI. | During Surgery
  Agreement of ICG and LSCI observations to determine flow in exposed vessels classified as no flow, delayed flow, or normal flow.

CONTACTS AND LOCATIONS:
Overall Officials: Michael T. Lawton, MD, Principal Investigator — Barrow Neurological Institute
Locations (1):
- Barrow Neurological Institute, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No